CLINICAL TRIAL: NCT00398580
Title: A Phase II, 28-Day, Randomized, Parallel-Group, Open-Label Study Evaluating the Efficacy and Safety of Twice Daily Oral Doses of Testosterone (150-400mg) Co-administered With 0.25mg Dutasteride Compared With 400mg Testosterone Alone and 0.25mg Dutasteride Alone in the Treatment of Hypogonadism
Brief Title: 28-Day Study of Testosterone Co-administered With Dutasteride in Hypogonadal Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDC106220
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hypogonadism; Hypogonadism, Male
Keywords: DHT; Testosterone; Hypogonadism; Dutasteride; Androgen deficiency
MeSH Terms: conditions — Hypogonadism; Eunuchism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nanomilled testosterone
Drug: Nanomilled dutasteride
Drug: commercially available dutasteride
  Other Names: Nanomilled testosterone; Nanomilled dutasteride

SUMMARY:
The combination of testosterone and dutasteride is intended for use in hypogonadal men. This study will evaluate the effect of 28-day repeat dosing of this combination with varying BID doses of testosterone (T), in combination with a fixed BID dose of dutasteride (D), as well as a testosterone alone arm, on T and D levels in the blood. The rationale is to look for the effects of each compound on the other, and to look for any safety problems that may result when the 2 drugs are given together.

ELIGIBILITY:
Inclusion criteria:

* Have a diagnosis of primary or secondary hypogonadism.
* Have very low testosterone levels on 2 separate days.
* Have a BMI within range of 18.5-35kg/m2.
* Have not taken dutasteride for one year, or finasteride for the past 3 months.

Exclusion criteria:

* Have had or have breast or prostate cancer, malabsorption syndrome, sleep apnea, psychiatric illness, polycythemia, or any other clinically significant current condition.
* Are diabetic with an HbA1c >= 8.
* Are taking any androgens, such as testosterone, saw palmetto.
* Are taking ritonavir, indinavir, itraconazole, ketoconazole, erythromycin, warfarin, digoxin, cholestyramine, or any dietary/herbal/vitamin supplements.
* Would donate more than 500 ML of blood over a 2 month period.
* Physician does not think it is a good idea for you to participate in the trial. - Are unwilling to abstain from alcohol during the study.
* Have a positive urine drug screen test.
* Plan to change your smoking habits during the course of the trial.
* Have Hepatitis C, Hepatitis B, or HIV.
* Have a lab or EKG abnormality.
* High or low blood pressure.
* Have used of any investigational drug or device during the study or within 30 days prior to 1st dosing of study medication.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety measured by: monitoring laboratory tests changes in blood pressure and heart rate and heart activity on an ECG machine | days 1 and 28

SECONDARY OUTCOMES:
Testosterone concentration . | on days 1 and 28
Pharmacokinetics of testosterone, DHT, estradiol, estrone & dutasteride | days 1 and 28.
Anabolic & androgenic Pharmacodynamic biomarkers | pre- and post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, M.D., Ph.D., FACP, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Seattle, Washington